CLINICAL TRIAL: NCT02397057
Title: A Double-Blinded, Multi-Center, Randomized, Placebo-Controlled Study to Investigate the Efficacy and Safety of Injectafer (Ferric Carboxymaltose) in the Treatment of Restless Legs Syndrome (RLS)
Brief Title: Placebo-Controlled Study to Investigate the Efficacy & Safety of Injectafer in the Treatment of RLS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1VIT14037
Record Dates: First submitted 2015-03-18; First posted 2015-03-24 (Estimated); Results first posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Restless Legs Syndrome (RLS)
MeSH Terms: conditions — Restless Legs Syndrome | interventions — ferric carboxymaltose; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Injectafer (Active Comparator): Two doses of Injectafer 750 mg undiluted dose at 100 mg/minute given 5 days apart for a total of 1500 mgs.
  Interventions: Drug: Injectafer
- Normal Saline (Placebo Comparator): IV Placebo (15ml of Normal Saline) IV push at 2ml/minute
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Injectafer
  Other Names: Ferinject®; Iroprem®; Renegy®
  Arms: Injectafer
Other: Placebo
  Other Names: Normal Saline
  Arms: Normal Saline

SUMMARY:
This will be a Phase III, double blinded, multi-center, randomized, placebo-controlled study. Eligible subjects will be randomized in a 1:1 ratio to receive Injectafer or Placebo on days 0 and 5. All treated subjects will be followed for efficacy and safety for 12 months. The subject's participation in the study will be for approximately 1 year from Day 0.

DETAILED DESCRIPTION:
This will be a Phase III, double blinded, multi-center, randomized, placebo-controlled study. Eligible subjects will be randomized in a 1:1 ratio to receive Injectafer or Placebo on days 0 and 5. All treated subjects will be followed for efficacy and safety for 12 months. Subjects will visit the clinic on Days 0 and 5 for treatment, and then on Days 14, 42, 168, and 365. In between the clinic visits subjects will be contacted remotely on Days 84, 126, 210, 252, 294, and 336. The subject's participation in the study will be for approximately 1 year from Day 0.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject's ≥18 years of age, willing and able to give informed consent to the study.
2. RLS symptoms affirming diagnosis. The IRLS Diagnostic Criteria must be met:

   1. An urge (distressing need) to move the legs usually associated with painful or uncomfortable sensations in the legs. The urge to move may be present without the uncomfortable sensations. The arms or other body parts may be involved in addition to the legs.
   2. The urge to move or unpleasant sensations are worse or exclusively present at rest or inactivity, such as lying down or sitting.
   3. The urge to move or unpleasant sensations are partially/temporarily relieved with walking or moving the legs.
   4. The urge to move or unpleasant sensations are worse in the evening or night than during the day or only occur in the evening or night. When symptoms are severe, the worsening at night may not be noticeable but must have been previously present.
3. Subjects should be on monotherapy for RLS. Treatment should be stable for at least 8 weeks prior to screening (See approved RLS Therapies/Regimen in Appendix III).
4. A score ≥15 on the IRLS Rating Scale at screening and on Day 0 prior to dosing.
5. Subjects on anti-depressants and sleep medications must be on a stable dose for at least 6 months.
6. Subject has regular sleep hours between 9 pm and 9 am.
7. Subjects at risk for pregnancy must have a negative pregnancy test at baseline and be practicing an acceptable form of birth control: have had a hysterectomy or tubal ligation, or otherwise be incapable of pregnancy, or have practiced any of the following methods of contraception for at least one month prior to study entry: hormonal contraceptives, spermicide with barrier, intrauterine device, or partner sterility.

Exclusion Criteria:

1. RLS 2° to other disease or injury.
2. Disorders that require treatment with the same medications used for RLS include: peripheral neuropathy and neurodegenerative disorders (i.e. Parkinson's Disease or Dementia).
3. Stage 4 - 5 CKD, subjects on dialysis or anticipated to start dialysis while participating in this study.
4. Any pain related (e.g., frequent muscle cramps, myalgia, fibromyalgia) or sleep related disorders (e.g. sleep apnea, unless on stable Continuous Positive Airway Pressure [CPAP]) which may confound the outcome measures.
5. Subjects with multiple sclerosis.
6. History of neuroleptic akathisia.
7. Parenteral iron use within 6 weeks prior to screening.
8. History of >10 blood transfusions in the past 2 years.
9. Anticipated need for blood transfusion during the study.
10. Known hypersensitivity reaction to any component of Injectafer® (Ferric Carboxymaltose).
11. Previously randomized to Injectafer® (FCM or VIT-45) in a clinical trial.
12. Current, active or acute or chronic infection other than viral upper respiratory tract infection
13. Malignancy (other than basal or squamous cell skin cancer or the subject has been cancer free for ≥ 5 years).
14. Pregnant or lactating women.
15. Seizure disorder currently being treated with medication.
16. Baseline ferritin ≥300 ng/mL.
17. Baseline TSAT ≥45%.
18. History of hemochromatosis, hemosiderosis, or other iron storage disorders.
19. AST or ALT greater than 2 times the upper limit of normal (ULN).
20. Hemoglobin greater than the ULN.
21. Known positive hepatitis B antigen (HBsAg), unless positive test can be attributed to receipt of hepatitis B vaccination in childhood or hepatitis C viral antibody (HCV) with evidence of active hepatitis (i.e., AST/ALT greater than the upper limit of normal).
22. Known positive HIV-1/HIV-2 antibodies (anti-HIV).
23. Received an investigational drug within 30 days before randomization.
24. Chronic alcohol or drug abuse within the past 6 months.
25. Any other pre-existing laboratory abnormality, medical condition or disease, which per the investigator may put the subject at risk if they participate in the study.
26. Subject unable or unwilling to comply with the study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Falone, MD, Study Director — American Regent, Inc.
Locations (19):
- United States (19):
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - Synergy San Diego, National City, California
  - Desert Valley Research, Rancho Mirage, California
  - Anderson Clinical Research, Redlands, California
  - Neurology Offices of South FL, Boca Raton, Florida
  - Elite Research Institute, Miami, Florida
  - MidAmmerica Neuroscience Institute, Lenexa, Kansas
  - Central Kentucky Research Assoc., Inc., Lexington, Kentucky
  - Neuromedical Clinical of Central Louisiana, Alexandria, Louisiana
  - Ctr for Brain & Neuro Care, LLC, Fulton, Maryland
  - Massachusetts General Hospital, Sleep Disorders Clinical Research Program, Boston, Massachusetts
  - Desert Neurology, Las Vegas, Nevada
  - Neurology Center of Las Vegas, Las Vegas, Nevada
  - Guilford Neurologic Associates, Greensboro, North Carolina
  - Metrolina Neurological Associates, Old Point Station, South Carolina
  - Saad Upstate Neurology, Spartanburg, South Carolina
  - Tri-State Mountain Neurology Associates, Johnson City, Tennessee
  - Egret Bay Neurology, Houston, Texas
  - The Polyclinic, Madison Center, Seattle, Washington

REFERENCES:
- [Derived] Earley CJ, Garcia-Borreguero D, Falone M, Winkelman JW. Clinical efficacy and safety of intravenous ferric carboxymaltose for treatment of restless legs syndrome: a multicenter, randomized, placebo-controlled clinical trial. Sleep. 2024 Jul 11;47(7):zsae095. doi: 10.1093/sleep/zsae095. PMID 38625730

RESULTS

PARTICIPANT FLOW:
Groups:
- Injectafer: Two doses of Injectafer 750 mg undiluted dose at 100 mg/minute given 5 days apart for a total of 1500 mgs.
  Injectafer
- Normal Saline: IV Placebo (15ml of Normal Saline) IV push at 2ml/minute
  Placebo
Period: Overall Study
Arm/Group | Injectafer | Normal Saline
Started | 105 (Two Normal Saline participants received "Injectafer". The data presented is considered accurate.) | 104
Completed | 94 | 91
Not Completed | 11 | 13
Not completed — Withdrawal by Subject | 6 | 7
Not completed — Lost to Follow-up | 4 | 3
Not completed — Death | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Subject did not receive study drug | 0 | 1

BASELINE CHARACTERISTICS:
Population: One subject did not receive study drug and was excluded from the Safety and Full Analysis Set Populations.
Groups:
- Total: Total of all reporting groups
Arm/Group | Injectafer | Normal Saline | Total
Number analyzed (Participants) | 105 | 103 | 208
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.3 (12.31) | 56.9 (13.73) | 57.6 (13.01)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One subject did not receive study drug and was excluded from the safety and full analysis population.
  Participants
    Female | 69 | 71 | 140
    Male | 36 | 32 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: One subject did not receive study drug and was excluded from the safety and full analysis population.
  Participants
    Hispanic or Latino | 12 | 9 | 21
    Not Hispanic or Latino | 93 | 94 | 187
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: One subject did not receive study drug and was excluded from the safety and full analysis population.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 1 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    Black or African American | 2 | 4 | 6
    White | 101 | 99 | 200
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 42 | 34 | 76
  Europe | 65 | 67 | 132
Height [Mean (Standard Deviation); unit: cm] | 167.6 (9.4) | 167 (9.4) | 167.3 (9.4)
Weight [Mean (Standard Deviation); unit: kg] | 82.8 (21.4) | 79.1 (20.8) | 81 (21.1)
Iron intolerance [Count of Participants; unit: Participants] — Population: One subject did not receive study drug and was excluded from the safety and full analysis population.
  Participants
    No | 104 | 103 | 207
    Yes | 1 | 0 | 1
RLS Medication-Related Augmentation [Count of Participants; unit: Participants] — Population: One participate did not receive study drug and was excluded from the safety and full analysis set population.
  Participants
    No augmentation | 51 | 53 | 104
    Uncertain augmentation | 31 | 33 | 64
    Definitive augmentation | 23 | 17 | 40

OUTCOME MEASURES:

1. Primary Outcome: International Restless Legs Syndrome (IRLS) Total Score Change From Baseline on Day 42
Description: Summary of the actual values of IRLS total score on baseline and Day 42, and the change from baseline to Day 42.
  Eligible subjects were to have met the following requirements prior to receiving additional treatment:
  A baseline score ≥ 15 on the International Restless Legs Syndrome (IRLS) Rating Scale. The minimum score is 15 with the maximum of 40. A score of less than 15 is not an indicator of RLS. However, a score of 15 or greater is an indicator of RLS. Further increase indicates more severe disease.
Time Frame: Baseline and Day 42
Population: One subject did not receive study drug and was excluded from the safety and Full analysis set population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Injectafer | Normal Saline
Number analyzed (Participants) | 105 | 103
score on a scale
  Baseline | 24.1 (6.27) | 24.5 (6.05)
  Day 42: number analyzed (Participants) | 87 | 69
  Day 42 | 15.6 (8.69) | 18.7 (8.94)
  Change from Baseline to Day 42 | -8.7 (8.44) | -5.9 (9.07)

2. Primary Outcome: Proportion of Patients Rated as Much or Very Much Improved With the Clinical Global Impression (CGI) Performed by Investigator (CGI-I)
Description: Responder is defined as subjects rated as much or very much improved with the CGI-I on Day 42. Summary of the number (percentage) of CGI-I responder. Per the protocol, the he CGI is a 3-item observer-rated scale that measures illness severity (CGIS), global improvement or change (CGIC) and therapeutic response. The scale requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention.
Time Frame: Day 42
Population: Responder(a), n/m(b) : a : Responder was defined as subjects rated as much or very much improved with the CGI-I.
  b : n is the number of responders; m is number of subjects who had non-missing results at the visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Injectafer | Normal Saline
Number analyzed (Participants) | 87 | 70
Participants | 38 | 25
Statistical Analysis 1: Comparison: Injectafer vs Normal Saline; Test type: Other — Observed cases, logistic regression analysis. Subjects with missing data on Day 42 were excluded from the statistical testing; p = 0.3690, Regression, Logistic — p-value was estimated by logistic regression with treatment, region (US, EUR), and baseline RLS medication-related augmentation as fixed factors, and baseline IRLS as a covariate; Odds Ratio (OR) = 1.35, 95% CI 2-sided [0.70 to 2.63]

3. Secondary Outcome: Clinical Global Impression-Improvement (CGI-S) by Subject
Description: Similar to the CGI-I except this is self-reported, 7-item scale for assessment of symptoms after treatment with the rating as: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.
Time Frame: Day 42
Population: Observed cases (n/m(a) [%])
  a: n is the number of subjects of the category, m is number of subjects who have non-missing results at the visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Injectafer | Normal Saline
Number analyzed (Participants) | 87 | 70
Participants
  Very much improved | 10 | 7
  Much improved | 30 | 19
  Minimal change | 31 | 16
  No Change | 10 | 12
  Minimally worse | 2 | 11
  Much worse | 3 | 4
  Very much worse | 1 | 1

4. Secondary Outcome: Restless Legs Syndrome Quality of Life (RLS-QLI) Change From Baseline to Day 42.
Description: The Restless Legs Syndrome Quality of Life (RLS-QLI) instrument, a self-assessment, 17-item questionnaire with four scales identified through factor analysis: Daily Function, Social Function, Sleep Quality, and Emotional Well-Being, developed to facilitate clinical research on RLS. Scoring Instructions below:
  1. Social Function = Sum (Items 1, 2, 3, 4), subtract 4, divide by 16, multiply by 100
  2. Daily Function = Sum (Items 5, 6, 13,14, 15, 16), subtract 6, divide by 24, multiply by 100
  3. Sleep Quality = Sum (Item 7, 8, 9, 17), subtract 4, divide by 18, multiply by 100
  4. Emotional Well-being = Sum (Items 10, 11, 12), subtract 3, divide by 12, multiply by 100
  Note: Resulting scores range between 0-100.
  Higher scores on the RLS-QLI indicate a lower quality of life. Lower scores indicate a higher quality of life.
Time Frame: Baseline and Day 42
Population: One subject did not receive study drug and was excluded from the Safety and Full Analysis Set Populations.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Injectafer | Normal Saline
Number analyzed (Participants) | 105 | 103
units on a scale
  Baseline | 55.6 (15.0) | 54.3 (13.08)
  Day 42: number analyzed (Participants) | 87 | 71
  Day 42 | 65.2 (15.49) | 62.8 (14.90)
  Change from Baseline to Day 42: number analyzed (Participants) | 87 | 71
  Change from Baseline to Day 42 | 9.0 (12.48) | 8.7 (14.61)

5. Secondary Outcome: Fatigue Linear Analog Scale Change From Baseline
Description: The Fatigue Linear Analog Scale is a self-assessment scale in which a 100 mm line is used to measure the severity of fatigue and its effect on a person's activities and lifestyle. The scale severity measure ranges from No Fatigue to Worst Possible Fatigue.
Time Frame: Baseline and Day 42
Population: One subject did not receive study drug and was excluded from the Safety and Full Analysis Set Populations.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Injectafer | Normal Saline
Number analyzed (Participants) | 104 | 103
units on a scale
  Baseline | 49.78 (26.32) | 57.34 (23.61)
  Day 42: number analyzed (Participants) | 84 | 69
  Day 42 | 38.90 (26.25) | 42.57 (27.13)
  Change from Baseline to Day 42: number analyzed (Participants) | 84 | 69
  Change from Baseline to Day 42 | -9.98 (27.55) | -16.50 (28.32)

6. Secondary Outcome: Medical Outcomes Study(MOS) Sleep Scale Change From Baseline to Day 42
Description: The MOS-Sleep scale, is a 12-item standardized, validated questionnaire for assessing sleep disturbance, sleep adequacy, somnolence, quantity of sleep, snoring, and awakening short of breath or with a headache which has been demonstrated to be sensitive to RLS treatment effects. This questionnaire provides information about sleep quality. Individual questions can be used for analysis but summary or index scores of a group of questions, is more commonly used in analysis.
  The "quantity of sleep" dimension is the average number of hours of sleep per night reported by the patient and the "optimal sleep" is a dichotomized version that is "yes" when the number of hours of sleep is 7 or 8. The scores of the dimensions and of the sleep problem index were converted to a 0 to 100 scale, with higher scores reflecting more of the attribute implied by the name (e.g. greater sleep disturbance, greater adequacy of sleep).
Time Frame: Change from Baseline and Day 42.
Population: Only participants with Sleep disturbance are included.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Injectafer | Normal Saline
Number analyzed (Participants) | 105 | 103
score on a scale | -13.086 (1.829) | -9.015 (1.902)
Statistical Analysis 1: Comparison: Injectafer vs Normal Saline; LOCF, ANCOVA Analysis; Test type: Other; p = 0.1108, ANCOVA; Least square(LS) mean difference = -4.071, 95% CI 2-sided [-9.083 to 0.941], Standard Error of Mean 2.542

7. Secondary Outcome: Time Off Pre-Enrollment Prescribed Restless Legs Syndrome (RLS) Medications
Description: Subjects could start tapering off pre-enrollment prescribed RLS medications after Day 5 until Day 365.
Time Frame: Time from Day 5 to Day 365
Population: Full Analysis Set Population. Subjects who discontinued or completed the study before an intervention were censored at the last study visit.
  Subjects Receiving RLS Intervention after Day 5.
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Injectafer | Normal Saline
Number analyzed (Participants) | 105 | 103
days | 34 [34 to 164] | 61 [61 to 183]
Statistical Analysis 1: Comparison: Injectafer vs Normal Saline; Test type: Other; p = 0.0002, Chi-squared, Corrected — p-value was estimated using continuity-corrected chi-square test

ADVERSE EVENTS:
Time Frame: 2 years, I month
Description: 209 participants were randomized of whom 208 received study drug: 105 who were randomized to Injectafer and 103 who were randomized to placebo. Two participants randomized to Placebo received Injectafer. Therefore the Numbers at Risk comprised 107 for Injectafer 101 for placebo.
Arm/Group | Injectafer | Normal Saline
All-Cause Mortality (participants affected / at risk) | 1/107 | 0/101
Serious Adverse Events (participants affected / at risk) | 6/107 | 4/101
Other Adverse Events (participants affected / at risk) | 72/107 | 19/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Injectafer (N=107) | Normal Saline (N=101)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colon cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Injectafer (N=107) | Normal Saline (N=101)
Nausea (Gastrointestinal disorders) | 10 (12) | 1 (1)
Feeling hot (General disorders) | 6 (6) | 0 (0)
Blood pressure increased (Investigations) | 5 (5) | 1 (1)
Alanine aminotransferase increased (Investigations) | 5 (5) | 1 (1)
Blood phosphorus decreased (Investigations) | 3 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 1 (1)
Blood pressure systolic increased (Investigations) | 5 (5) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 8 (9) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Dizziness (Nervous system disorders) | 8 (8) | 1 (1)
Headache (Nervous system disorders) | 5 (5) | 6 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hot flush (Vascular disorders) | 5 (5) | 1 (1)
Flushing (Vascular disorders) | 6 (6) | 0 (0)
Gamma-Glutamyl Transferase Increase (Investigations) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2016-06-02): https://cdn.clinicaltrials.gov/large-docs/57/NCT02397057/Prot_000.pdf
  • Statistical Analysis Plan (2016-11-22): https://cdn.clinicaltrials.gov/large-docs/57/NCT02397057/SAP_001.pdf